CLINICAL TRIAL: NCT02195609
Title: Randomized Open Label Study to Evaluate the Effect of (Omega-3) EPA + Docosahexaenoic Acid (DHA) vs Soy Isoflavones in 100 Postmenopausal Women Between 45-65 Years With Moderate to Severe Vasomotor Symptoms.
Brief Title: Evaluate the Effect of Omega-3 vs Soy Isoflavones in Postmenopausal Women With Moderate to Severe Vasomotor Symptoms
Acronym: OMEGASI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Palacios (Other)
Collaborators: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IP-2013-01
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Menopause; Hot Flashes
Keywords: Vasomotor Symptoms Associated With Menopause; Menopause; Hot Flashes; Postmenopausal Women
MeSH Terms: conditions — Hot Flashes | interventions — Docosahexaenoic Acids; Soybean Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 (Other): 600 mg (EPA, DHA and Omega-3) twice a day
  Interventions: Dietary Supplement: Omega-3
- Soy Isoflavones (Other): 54.4mg oral twice a day
  Interventions: Dietary Supplement: Soy Isoflavones

INTERVENTIONS:
Dietary Supplement: Omega-3 — 600 mg oral twice a day
  Other Names: Om3gafort
  Arms: Omega-3
Dietary Supplement: Soy Isoflavones — 54.4 mg oral twice a day
  Other Names: Flavia
  Arms: Soy Isoflavones

SUMMARY:
This study is aiming to evaluate changes in vasomotor symptoms in postmenopausal women treated for 4 months with Omega-3 vs Soy Isoflavones.

DETAILED DESCRIPTION:
This is a non-inferiority study of Omega 3 versus Soy Isoflavones, being each patient its own control from the baseline.

In order to determine the difference observed in the evolution of intensity, frequency and the total number of hot flashes in 4 months in patients treated with Omega-3 vs Soy Isoflavones, is planned to include at least 100 patients, 50 per treatment arm.

It si estimated a standar deviation of 0.5%, and a 10% lost follow-up rate.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory and can complete all study procedures, which are able to read, understand and sign an informed consent and willing to come to the center for study visits.
* Postmenopausal (≥ 1 year of amenorrhea) or 6 months or more of amenorrhea with follicle stimulating hormone (FSH) ≥ 40 IU / L.
* BMI ≥ 18 kg/m2 and ≤ 30 kg/m2
* Flushing of moderate to severe intensity.

Exclusion Criteria:

* Women with surgical menopause.
* Treatment with hormone replacement therapy (HRT) in the 3 months prior to inclusion
* Uterine bleeding after menopause with undetermined cause in the 12 months prior to screening.
* Presence or history of malignancy in the past 5 years.
* Malabsorption syndrome.
* Hype or uncontrolled hypothyroidism.
* Dyslipidemia (LDL-cholesterol> 189 mg / dl or medical criteria) requiring an specific treatment of proven effectiveness.
* Chronic renal disease.
* Uncontrolled or untreated hypertension.
* Treatment with isoflavones, tibolone, Selective Estrogen Receptors Moderators (SERM´s) in the past 3 months prior to the testing selection period.
* Hormonal treatment with androgens, estrogens, progestins, alone or combined oral, transdermal, vaginal (including promestriene) or implant, in the last 3 months prior to testing selection period.
* Patients who receive or require treatment with antidepressants or anticonvulsants
* Patients with mental illness.
* History of noncompliance with taking medication.
* Suspected or abuse of alcohol or other drugs during the 12 months preceding the selection.
* Use of any experimental drug or device within 30 days prior to the selection.
* Any other condition or finding that a judgment of the investigator may jeopardise the tral conduct according to the protocol.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the changes in vasomotor symptoms. | 0 to 4 months
  To evaluate the changes in vasomotor symptoms in postmenopausal women measured by a hot flushes self-completed diary .

SECONDARY OUTCOMES:
Cardiovascular risk factors | 0 and 4 months
  serum cholesterol
Satisfaction with treatment | at month 1 and 4
  Treatment Satisfaction Questionnaire for Medication
Mood status | 0, 1 and 4 months
  Hospital Anxiety and Depression Scale (HADS)
General health status | months 0, 1 and 4
  General health status by Short-Form 36 (SF-36) questionnaire
Rating memory status | at 0, 1 and 4 months
  Alteration of the memory test (T@M)
Cardiovascular risk factors | 0 amd 4 months
  serum triglycerides
Cardiovascular risk factors | 0, 1 and 4 months
  Blood pressure
Cardiovascular risk factors | 0, 1 and 4 months
  Body mass index
Cardiovascular risk factors | 0, 1 and 4 months
  abdominal circumference

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Palacios, MD, Study Director — President of the European Foundation Woman and Health,Past President and Honorary Member of the Spanish Menopause Society, President of the Council of Affiliated Menopause Societies (CAMS)
Locations (1):
- Instituto Palacios, Madrid, Madrid, Spain